CLINICAL TRIAL: NCT03498716
Title: A Phase III, Multicenter, Randomized, Open-Label Study Comparing Atezolizumab (Anti PD-L1 Antibody) in Combination With Adjuvant Anthracycline/Taxane-Based Chemotherapy Versus Chemotherapy Alone in Patients With Operable Triple Negative Breast Cancer
Brief Title: A Study Comparing Atezolizumab (Anti PD-L1 Antibody) In Combination With Adjuvant Anthracycline/Taxane-Based Chemotherapy Versus Chemotherapy Alone In Patients With Operable Triple-Negative Breast Cancer
Acronym: IMpassion030
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by the sponsor following interim analysis as the primary endpoint of iDFS crossed the pre-specified futility boundary of hazard ratio > 1 in the Intent-to-Treat (ITT) population.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Breast International Group (Other); Alliance Foundation Trials, LLC. (Other); Jules Bordet Institute (Other); Frontier Science & Technology Research Foundation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO39391; 2016-003695-47 (EudraCT Number); BIG 16-05 (Other: Breast International Group (BIG)); AFT-27 (Other: Alliance Foundation Trials); ALEXANDRA (Other: Breast International Group (BIG))
Record Dates: First submitted 2018-02-28; First posted 2018-04-17 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Paclitaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Chemotherapy (Experimental): Participants will receive atezolizumab (in combination with chemotherapy as described below) every 2 weeks for 10 doses, followed by atezolizumab maintenance therapy every 3 weeks to complete 1 year of treatment from the first dose
  Chemotherapy will consist of paclitaxel every week for 12 weeks, followed by dose-dense doxorubicin +cyclophosphamide or dose-dense epirubicin + cyclophosphamide every 2 weeks, for 4 doses supported with Granulocyte Colony-Stimulating Factor (G-CSF) or Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF)
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Dose-dense Doxorubicin or dose-dense Epirubicin; Drug: Cyclophosphamide
- Chemotherapy (Active Comparator): Chemotherapy will consist of paclitaxel every week for 12 weeks, followed by dose-dense doxorubicin +cyclophosphamide or dose-dense epirubicin + cyclophosphamide every 2 weeks, for 4 doses supported with Granulocyte Colony-Stimulating Factor (G-CSF) or Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF)
  Interventions: Drug: Paclitaxel; Drug: Dose-dense Doxorubicin or dose-dense Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV, 840 mg every 2 weeks, for 10 doses.
  Atezolizumab maintenance will be administered by IV, 1200 mg every 3 weeks to complete 1 year
  Arms: Atezolizumab + Chemotherapy
Drug: Paclitaxel — Paclitaxel will be administered by IV, 80 mg/m^2 every week for 12 weeks.
Drug: Dose-dense Doxorubicin or dose-dense Epirubicin — Dose-dense doxorubicin will be administered by IV, 60 mg/m^2 every 2 weeks for a total of 4 doses.
  Or
  Dose-dense epirubicin will be administered by IV, (90 mg/m^2) every 2 weeks for a total of 4 doses
Drug: Cyclophosphamide — Cyclophosphamide will be administered by IV, 600 mg/m^2 every 2 weeks for 4 doses

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of adjuvant atezolizumab in combination with paclitaxel, followed by atezolizumab, dose-dense doxorubicin or epirubicin (investigator's choice), and cyclophosphamide, compared with paclitaxel followed by dose-dense doxorubicin or epirubicin (investigator's choice) and cyclophosphamide alone in patients with Stage II-III TNBC (Triple Negative Breast Cancer)

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic operable Stage II-III breast cancer
* Histologically documented TNBC (Triple Negative Breast Cancer)
* Confirmed tumor PD-L1 evaluation as documented through central testing of a representative tumor tissue specimen
* Adequately excised: Patients must have undergone either breast-conserving surgery or mastectomy/nipple- or skin-sparing mastectomy
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm.
* No more than 8 weeks (56 days) may elapse between definitive breast surgery and randomization.
* Representative formalin-fixed, paraffin embedded (FFPE) tumor specimen from surgical resection in paraffin blocks (preferred) or at least 25 unstained slides.

Exclusion Criteria

* Prior history of invasive breast cancer
* For the currently diagnosed breast cancer, any previous systemic anti-cancer treatment (e.g., neoadjuvant or adjuvant), including, but not limited to, chemotherapy, anti-HER2 therapy.
* Previous therapy with anthracyclines or taxanes for any malignancy
* Cardiopulmonary dysfunction
* Prior malignancies within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Urinary outflow obstruction
* Active tuberculosis
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during study treatment or within 5 months following the last dose of Atezolizumab (for patients randomized to Atezolizumab)
* Prior allogeneic stem cell or solid organ transplant
* Treatment with systemic immunosuppressive medications within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressive medication during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2199 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (364):
- United States (17):
  - John Muir Health Clinical Research Center, Concord, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Martin-O?Neil Cancer Center, St. Helena, California
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Advocate Illinois Masonic Outpatient Center for Advanced Care, Chicago, Illinois
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Fairview Southdale Medical Oncology Clinic, Edina, Minnesota
  - HCA Midwest Division, Kansas City, Missouri
  - New Hampshire Hematology Oncology, Manchester, New Hampshire
  - Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Rochester General Hospital; Lipson Cancer and Blood Center, Rochester, New York
  - SCRI, Nashville, Tennessee
  - Intermountain Precision Genomics Cancer Research Clinic-Dixie, St. George, Utah
  - St. Mary's Medical Center, Huntington, West Virginia
- Argentina (9):
  - Centro de Oncologia e; Investigacion Buenos Aires - COIBA, Berazategui
  - INSTITUTO DE INVESTIGACIONES METABOLICAS (IDIM); Oncology, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Instituto de Oncología de Rosario, Rosario
  - Centro Medico San Roque, San Miguel de Tucumán
  - Fundación Ars Medica, San Salvador de Jujuy
  - Centro de Investigacion Clinica - Clinica Viedma S.A.; Oncology Department, Viedma
- Australia (15):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Icon Cancer Foundation; Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Mater Hospital; Cancer Services, South Brisbane, Queensland
  - Icon Cancer Foundation; Icon Cancer Care Southport, Southport, Queensland
  - Princess Alexandra Hospital; Cancer Trials Unit, Woolloongabba, Queensland
  - Royal Adelaide Hospital; Cancer Centre, Adelaide, South Australia
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital Olivia Newton John Cancer Centre, Heidelberg, Victoria
  - Maroondah Hospital; Breast Clinic, Ringwood East, Victoria
- Austria (7):
  - Medical University Innsbruck; Frauenklinik Innsbruck, Dept Gyn, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern; Interne 1 - Hämato-Onkologie, Linz
  - Uniklinikum Salzburg, LKH; Univ.Klinik f. Innere Medizin III der PMU, Salzburg
  - AKH - Medizinische Universität Wien; Department of Oncology, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Salzkammergut-Klinikum Voecklabruck, Vöcklabruck
  - Klinikum Kreuzschwestern Wels; Iv. Interne Abt., Wels
- Belgium (8):
  - AZ KLINA, Brasschaat
  - Institut Jules Bordet, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHC MontLégia, Liège
  - Chr de La Citadelle, Liège
  - CHU Ambroise Paré, Mons
  - Clinique Sainte-Elisabeth; Oncologie, Namur
  - Vitaz, Sint-Niklaas
- Brazil (14):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Jardim Amália, Volta Redonda, Rio de Janeiro
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Instituto Do Câncer Do Estado de São Paulo Octávio Frias de Oliveira, São Paulo, São Paulo
  - Instituto Brasileiro de Controle Do Câncer ? São Camilo Oncologia, São Paulo, São Paulo
- China (28):
  - Peking University People's Hospital, Beijing
  - Beijing Hospital; Internal Medicine-Oncology, Beijing
  - Beijing Union Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun yat-sen University Cancer Center; Internal Medicine of Oncology, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Sun Yat-Sen University Cancer Center - Huangpu Campus, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Luoyang Central Hospital, Luoyang
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - The University of Hong Kong-Shenzhen Hospital; Local Ethic Committee, Shenzhen
  - Hebei Medical University Fourth Hospital;(Tumor Hospital of Hebei Province), Shijiazhuang
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Nemocnice Horovice, NH Hospital a.s.; Oncology Department, Hořovice
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Krajska nemocnice T. Bati, a.s., Zlín
- Denmark (3):
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling, Klinisk Forsknings Enhed, Odense C
  - Sygehus Lillebælt, Vejle, Vejle
- France (35):
  - Centre Hospitalier Regional Metz-Thionville - Hopital de Mercy, Ars-Laquenexy
  - Institut Sainte Catherine, Avignon
  - CH de Beauvais, Beauvais
  - CHU Jean Minjoz, Besançon
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - CHRU De Brest - Hopital Morvan - Institut De Cancerologie Et D'Hematologie, Brest
  - CRLCC-Francois Baclesse; Oncologie Médicale, Caen
  - CH de Cholet; oncologie, Cholet
  - Centre Hospitalier de Compiegne, Compiègne
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Clinique Chenieux; Oncology, Limoges
  - Centre Hospitalier Bretagne Sud, Lorient
  - Hopital Prive Jean Mermoz, Lyon
  - Hôpital Saint Joseph, Marseille
  - Clinique Clémentville, Montpellier
  - Institut régional du Cancer Montpellier, Montpellier
  - l'Hôpital privé du Confluent SAS, Nantes
  - Centre Antoine Lacassagne, Nice
  - CH Annecy Genevois site Annecy; Oncologie, Pringy
  - Chi De Cornouaille; Oncologie Hospitalisation, Quimper
  - Institut Jean Godinot, Reims
  - Institut du Cancer Coulancy Reims, Reims
  - Centre Henri Becquerel, Rouen
  - Institut De Cancerologie Lucien Newrth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Du Leman - Site Georges Pianta, Thonon-les-Bains
  - Institut Claudius Régaud, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Hopital Prive Drome Ardeche; Hopital De Jour, Valence
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Germany (26):
  - Studienzentrum Berlin City, Berlin
  - St. Elisabeth-Krankenhaus, Cologne
  - St. Johannes-Hospital, Dortmund
  - Onkozentrum Dres. Göhler, Dresden
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Praxis für Hamatologie und Onkologie, Erfurt
  - Onkodok GmbH, Gütersloh
  - Albertinen-Krankenhaus Klinik f.Gynäkologie und Geburtshilfe, Hamburg
  - Ärztehaus am Bahnhofsplatz; Praxis Uleer/Pourfard, Hildesheim
  - ViDia Christliche Kliniken Karlsruhe, Vincentius-Diakonissen-Kliniken gAG; Frauenklinik, Karlsruhe
  - Klinikum Ludwigsburg; Studiensekretariat, Ludwigsburg
  - St. Vincenz-Elisabeth-Hospital; Katholisches Klinikum Mainz, Mainz
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Dres. Michael Maasberg Marion Schmitz und Maria Theresia Keller, Mayen
  - Klinikum Memmingen; Abt.Gynäkologie, Memmingen
  - Johannes Wesling Klinikum Minden; Hämatologie, Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Brustzentrum Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - Klinikum der Universität München; Frauenklinik - Onkologie II, München
  - Klinikum Neumarkt; Frauenklinik, Neumarkt in der Oberpfalz
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Johanniter Frauenklinik Stendal Germany, Stendal
  - Gynäkologie Kompetenzzentrum; Praxis Dr. med. Carsten Hielscher, Stralsund
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
  - GRN-Klinik Weinheim; Abt.Gynäkologie und Geburtshilfe, Weinheim
  - Marien-Hospital Witten, MVZ Witten, Witten
  - Klinikum Worms; Frauenklinik; Klinik für Gynäkologie und Geburtshilfe, Worms
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital; Clinical Oncology, Hong Kong
  - Queen Elizabeth Hospital Department of Clinical Oncology, Kowloon
- Hungary (3):
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Pécsi Tudományegyetem; Klinikai Központ Onkoterápiás Intézet, Pécs
- Ireland (2):
  - Mater Misecordiae University Hospital, Dublin
  - Beaumont Hospital; Cancer Clinical Trials Unit, Dublin
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Med Org Kiryat; Oncology Institute, Jerusalem
  - Meir Medical center, Pediatrics, Kfar Saba
  - Rabin MC; Davidof Center - Oncology Institute, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (22):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Abruzzo
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S.Orsola Malpighi; UO Farmacia Clinica, Bologna, Emilia-Romagna
  - U.O Medicina Oncologica Ospedale di Carpi, Carpi, Emilia-Romagna
  - Ospedale Degli Infermi - Faenza; Oncologia Medica, Faenza, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Ospedale degli Infermi, Rimini, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia, Udine, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Azienda Ospedaliero Universitaria San Martino, Genoa, Liguria
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - Ospedale Mater Salutis, Legnago (VR), Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Salvatore Maugeri, Pavia, Lombardy
  - Policlinico San Mattea, Pavia, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria, Piedmont
  - Ospedale Degli Infermi Di Biella; Reparto Oncologia Medica, Ponderano (BI), Piedmont
  - Ospedale Santa Maria Annunziata; Oncologia, Bagno a Ripoli, Tuscany
  - Azienda Usl 7; Dept. Oncologico, Poggibonsi, Tuscany
  - Nuovo Ospedale Di Prato, Prato, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia, Umbria
- Japan (22):
  - Aichi Cancer Center Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Fukushima Medical University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Naha-nishi Clinic, Okinawa
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - St. Luke's Internat. Hospital, Breast Surgical Oncology, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Mexico (9):
  - Iem-Fucam, D.F., Mexico CITY (federal District)
  - Instituto Nacional De Cancerologia; Oncology; Tumores Mamarios, Distrito Federal, Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - Merida | Investigacion Clinica, Mérida, Yucatán
  - CENEIT Oncologicos; DENTRO DE CONDOMINIO SAN FRANCISCO, Mexico City
  - Centro Medico Dalinde, Mexico City
- Peru (3):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud; Oncology & Haemathology, Arequipa
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Oncosalud Sac; Oncología, Lima
- Poland (4):
  - Instytut MSF Sp. z o.o., ?ód?
  - MedPolonia, Poznan
  - Wielkopolskie Centrum Onkologi, Poznan
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy; Klinika Onkologii, Warsaw
- Romania (3):
  - "Filantropia" Clinical Hospital; Gynecological Oncology, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca; Oncologie Medicala, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
- Russia (27):
  - Medsi Clinic, Moscow, Adygeya Republic
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - Oncologica Dispensary #2, Sochi, Krasnodarskiy Kray
  - Evimed, Chelyabinsk, Kurgan Oblast
  - Moscow Clinical Scientific Center, Moscow, Moscow Oblast
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
  - Nizhny Novgorod Regional Clinical Oncology Center, Nizhny Novgorod, Niznij Novgorod
  - Mordovia State University, Saransk, Respublika Mordoviya
  - National Medical Research Center for Oncology, Rostov-on-Don, Rostov Oblast
  - LLC Strategic Medical Systems, Saint Petersburg, Sankt-Peterburg
  - EosMed LLC, Saint Petersburg, Sankt-Peterburg
  - Private Healthcare Institution Clinical Hospital RZhD Medicine, Saint Petersburg, Sankt-Peterburg
  - LCC Center of Palliative Medicine - Devita, Saint Petersburg, Sankt-Peterburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg, Sankt-Peterburg
  - Pyatigorsky Oncologic Dispensary, Pyatigorsk, Stavropol Kray
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - Regional Oncology Hospital, Irkutsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Regional Oncology Dispensary; Dept of Chemotherapy, Novgorod Veliky
  - BIH at Omsk Region "Clinical Oncology Dispensary", Outpatient clinic, Omsk
  - Multidisciplinary clinic Reaviz, Samara
  - Samara Regional Oncology Dispensary, Samara
  - Regional Clinical Hospital, Saratov
  - SHI Volgograd Regional Clinical Oncological Dispensary#1, Volgograd
- Singapore (2):
  - National University Hospital; Medical Oncology, Singapore
  - National Cancer Centre, Singapore
- South Korea (17):
  - Chungbuk National University Hospital, Cheongju-si
  - Soon Chun Hyang University Cheonan Hospital, Dongnam-gu, Cheonan-si
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital; Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hosiptal, Ulsan
  - Wonju Christian Hospital, Wŏnju
- Spain (30):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital General De Catalunya; Servicio de Oncologia, Sant Cugat del Vallès, Barcelona
  - Consorci Hospitalari de Terrassa, Terrassa, Barcelona
  - Hospital de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Provincial Castellón, Castellon de LA Plana/castello de LA Plana, Castellon
  - Centro Oncologico de Galicia COG; Medical Oncology, A Coruña, LA Coruña
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Infanta Sofia; Servico de Oncologia, San Sebastián de los Reyes, Madrid
  - Complexo Hospitalario de Vigo. Hospital Álvaro Cunqueiro; Servicio de Oncología, Vigo, Pontevedra
  - Hospital Universitari Sant Joan de Reus; Planta baja, color lila, Reus, Tarragona
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Complejo Hospitalario de Jaen, Jaén
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncológico Clara Campal Ensayos Clínicos START, Madrid
  - Hosp Univ Fundacion Alcorcon, Madrid
  - Hospital Universitario de Fuenlabrada; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Quirón Sagrado Corazón, Seville
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
- Switzerland (3):
  - Hirslanden Medical Center - Tumorzentrum, Aarau
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - Brust-Zentrum Zürich AG Seefeldstrasse 214 Zürich, Zurich
- Taiwan (10):
  - Chunghua Christian hospital, Changhua
  - Kaohsiung Medical University Hospital; Chung-Ho Memorial Hospital, Kaoshiung City
  - E-Da Cancer Hospital; Hematology- Oncology Department, Kaoshiung
  - Chi Mei Medical Center Liou Ying Campus, Liuying Township
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital - Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- Thailand (7):
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Ramathibodi Hospital; Medicine/Oncology, Bangkok
  - Siriraj Hospital; Clinical Research Center, Pharmacy Department, Bangkok
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Lampang Cancer Hospital, Lampang
  - King Chulalongkorn Memorial Hospital; Faculty of Medicine Chulalongkorn University, Patumwan
- Turkey (Türkiye) (5):
  - Baskent Universitesi Adana Dr. Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Uludag Universitesi - Saglik Uygulama ve Arastirrma Merkezi, Bursa
  - Izmir Ekonomi Universitesi Medical Park Hastanesi, Izmir
  - Mersin Universitesi Tip Fakultesi Hastanesi; Tibbi Onkoloji Birimi, Mersin
  - Medikal Park Samsun, Samsun
- Ukraine (16):
  - Yulis Medical and Diagnostic Center, Zaporizhzhia, Katerynoslav Governorate
  - MI "Clinical Oncological Dispensary" of Dnipro Reg Council; chemotherapy department, Dnipro, KIEV Governorate
  - Municipal Institution Odesa Regional Oncology Dispensary, Odesa, KIEV Governorate
  - Vinnytsya Regional Clinical Oncology Dispensary, Vinnytsia, Podolia Governorate
  - Regional Oncology Center; Department of Mammology, Chernihiv
  - Chernivtsi Regional Clinical Oncology Dispensary, Chernivtsi
  - City Clinical Hospital #4, Dnipropetrovsk
  - Municipal Institution Kirovograd Regional Oncology Dispensary, Kirovograd
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council; Chemotherapy Department, Kryvyi Rih
  - Volyn Regional Oncology Dispensary, Lutsk
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Sumy Reg. Clin. Oncological Dispensary; Thoracall Department, Sumy
  - CCCH City Oncological Center SHEI Uzhgorod NU, Uzhhorod
  - Transkarpathian Regional Oncology Clinic; Chemotherapy, Uzhhorod
  - Zaporizhzhia Regional Clinical Oncology Dispensary; Zaporizhzhya State Medical University, Zaporizhzhya
- United Kingdom (6):
  - NHS Lothian - Western General Hospital; NHS Lothian - Western General Hospital, Edinburgh
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - Leeds Teaching Hosp NHS Trust;St James's Institute of Onc, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - University Hospitals of North Midlands NHS Trust-Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Ignatiadis M, Bailey A, McArthur H, El-Abed S, de Azambuja E, Metzger O, Chui SY, Dieterich M, Perretti T, Shearer-Kang E, Molinero L, Steger GG, Jassem J, Lee SC, Higgins M, Zarba J, Schmidt M, Gomez H, Guerrero Zotano A, Moscetti L, Chiu J, Munzone E, Ben-Baruch NE, Bajetta E, Ohno S, Im SA, Werutsky G, Gal-Yam EN, Gonzalez Farre X, Tseng LM, Jacot W, Gluz O, Shao Z, Shparyk Y, Zimina A, Winer E, Cameron DA, Viale G, Saji S, Gelber R, Piccart M. Adjuvant Atezolizumab for Early Triple-Negative Breast Cancer: The ALEXANDRA/IMpassion030 Randomized Clinical Trial. JAMA. 2025 Jan 30;333(13):1150-60. doi: 10.1001/jama.2024.26886. Online ahead of print. PMID 39883436
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed Stage II-III primary invasive Breast cancer (BC) that is of triple negative phenotype and who were to be treated with adjuvant systemic chemotherapy following definitive surgery, were enrolled in 342 centers in 31 countries.
Pre-assignment Details: A total of 2199 participants were enrolled in the study. Participants were randomized in a 1:1 ratio to receive Atezolizumab and Chemotherapy or Chemotherapy alone.
Groups:
- Chemotherapy: Participants were administered paclitaxel, 80 milligram per square meter (mg/m^2), intravenous (IV) infusion weekly (QW) for maximum of 36 weeks followed by dose-dense doxorubicin, 60 mg/m^2 or dose-dense epirubicin, 90 mg/m^2 IV (investigator's choice) plus cyclophosphamide, 600 mg/m^2, IV repeated every 2 weeks (Q2W) for a maximum of 20 weeks supported with granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) treatment.
- Atezolizumab and Chemotherapy: Participants were administered atezolizumab 840 mg, IV infusion, Q2W in combination with chemotherapy (paclitaxel 80 mg/m^2, IV infusion QW for maximum of 22 weeks followed by dose-dense doxorubicin, 60 mg/m^2 or dose-dense epirubicin, 90 mg/m^2, IV (investigator's choice) plus cyclophosphamide, 600 mg/m^2, IV repeated Q2W for maximum of 17 weeks supported with G-CSF or GM-CSF treatment followed by atezolizumab, 1200 mg IV infusion every 3 weeks (Q3W) as a maintenance therapy to complete 1 year of atezolizumab treatment from the first dose.
Period: Overall Study
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Started | 1098 | 1101
Safety Evaluable Population (Safety Evaluable Population included all participants who received any amount of any study drug.) | 1084 | 1093
Completed | 0 | 0
Not Completed | 1098 | 1101
Not completed — Withdrawal by Subject | 88 | 73
Not completed — Study Terminated By Sponsor | 933 | 927
Not completed — Lost to Follow-up | 15 | 26
Not completed — Disease Relapse | 0 | 1
Not completed — Death | 58 | 72
Not completed — Physician Decision | 4 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants, whether or not the assigned study treatment was received.
Groups:
- Chemotherapy: Participants were administered paclitaxel, 80 mg/m^2, IV infusion QW for maximum of 36 weeks followed by dose-dense doxorubicin, 60 mg/m^2 or dose-dense epirubicin, 90 mg/m^2 IV (investigator's choice) plus cyclophosphamide, 600 mg/m^2, IV repeated every Q2W for a maximum of 20 weeks supported with G-CSF or GM-CSF treatment.
- Atezolizumab and Chemotherapy: Participants were administered atezolizumab 840 mg, IV infusion, Q2W in combination with chemotherapy (paclitaxel 80 mg/m^2, IV infusion QW for maximum of 22 weeks followed by dose-dense doxorubicin, 60 mg/m^2 or dose-dense epirubicin, 90 mg/m^2, IV (investigator's choice) plus cyclophosphamide, 600 mg/m^2, IV repeated Q2W for maximum of 17 weeks supported with G-CSF or GM-CSF treatment followed by atezolizumab, 1200 mg IV infusion every Q3W as a maintenance therapy to complete 1 year of atezolizumab treatment from the first dose.
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy | Total
Number analyzed (Participants) | 1098 | 1101 | 2199
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (11.4) | 52.3 (11.9) | 52.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1094 | 1101 | 2195
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 75 | 175
  Not Hispanic or Latino | 906 | 950 | 1856
  Unknown or Not Reported | 92 | 76 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 29 | 57
  Asian | 401 | 423 | 824
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 8 | 10
  White | 567 | 554 | 1121
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 99 | 86 | 185

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-Free Survival (iDFS)
Description: iDFS was defined as the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer involving the same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive breast cancer recurrence (an invasive breast cancer in the axilla, regional lymph nodes, chest wall, &/or skin of the ipsilateral breast); Ipsilateral second primary invasive breast cancer; Contralateral invasive breast cancer; Distant recurrence (evidence of breast cancer in any anatomic site [other than the sites mentioned]) that has either been histologically confirmed &/or clinically/radiographically diagnosed as recurrent invasive breast cancer; & Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: From randomization until the occurrence of an iDFS event or death from any cause, whichever occurred earlier (up to 5 years)
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred. | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred.
Statistical Analysis 1: Comparison: Chemotherapy vs Atezolizumab and Chemotherapy; Test type: Superiority — Stratified Analysis: The stratification factors used in the analysis are axillary nodal status, surgery (breast conserving vs. mastectomy),and tumor PD-L1 status; p = 0.3846, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.87 to 1.42]

2. Secondary Outcome: Invasive Disease-Free Survival (iDFS) in the Subpopulation With Programmed Death-ligand 1 (PD-L1) Selected Tumor Status (IC1/2/3)
Description: iDFS = the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer involving the same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive breast cancer recurrence (an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); Ipsilateral second primary invasive breast cancer, Contralateral invasive breast cancer, Distant recurrence (i.e., evidence of breast cancer in any anatomic site [other than the sites mentioned]) that has either been histologically confirmed and/or clinically/radiographically diagnosed as recurrent invasive breast cancer and Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: as for outcome 1
Population: PD-L1-positive subpopulation included participants in the ITT population whose PD-L1 status was IC1/2/3 at the time of randomization. ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 782 | 785
months | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred. | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred.

3. Secondary Outcome: Invasive Disease-Free Survival (iDFS) in the Node Positive Subpopulation
Description: iDFS = the time from randomization until the date of the first occurrence of one of the following events: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer involving the same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive breast cancer recurrence (an invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); Ipsilateral second primary invasive breast cancer; Contralateral invasive breast cancer; Distant recurrence (evidence of breast cancer in any anatomic site [other than the sites mentioned]) that has either been histologically confirmed and/or clinically/radiographically diagnosed as recurrent invasive breast cancer; and Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: as for outcome 1
Population: Node positive subpopulation included all participants in the ITT population whose lymph node (LN) status was positive at the time of randomization. ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 533 | 534
months | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred. | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from randomization to the date of death due to any cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: From randomization up to death from any cause (up to 5 years)
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for OS were not estimable due to too few events having occurred. | NA [NA to NA] — Median and 95% CI for OS were not estimable due to too few events having occurred.

5. Secondary Outcome: Invasive Disease-Free Survival (iDFS) Including Second Primary Non-Breast Invasive Cancer
Description: iDFS = the time from randomization until the date of first occurrence of one of the events: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer involving same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive breast cancer recurrence (an invasive breast cancer in axilla, regional lymph nodes, chest wall, &/or skin of the ipsilateral breast); Ipsilateral second primary invasive breast cancer; Second primary non-breast invasive cancer; Contralateral invasive breast cancer; Distant recurrence (i.e., evidence of breast cancer in any anatomic site [other than sites mentioned]) that has either been histologically confirmed &/or clinically/radiographically diagnosed as recurrent invasive breast cancer; Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: From randomization up to death from any cause (up to 5 years)
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred | NA [NA to NA] — Median and 95% CI for iDFS were not estimable due to too few events having occurred

6. Secondary Outcome: Recurrence-Free Interval (RFI)
Description: Recurrence-Free Interval (RFI) was defined as the time from randomization to the first occurrence of any recurrence (local, regional [including invasive ipsilateral tumor and invasive locoregional tumor], or distant), as determined by investigators. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis, participants with no events who died, or participants with no post-baseline information were censored.
Time Frame: From randomization up to 5 years
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for RFI were not estimable due to too few events having occurred | NA [NA to NA] — Median and 95% CI for RFI were not estimable due to too few events having occurred

7. Secondary Outcome: Distant Recurrence-Free Interval (DRFI)
Description: Distant Recurrence-Free Interval (DRFI) was defined as the time from randomization to the distant breast cancer recurrence. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis, participants with no events who died, or participants with no post-baseline information were censored.
Time Frame: From randomization up to 5 years
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for DRFI were not estimable due to too few events having occurred | NA [NA to NA] — Median and 95% CI for DRFI were not estimable due to too few events having occurred

8. Secondary Outcome: Disease-Free Survival (DFS)
Description: Disease-Free Survival (DFS) was defined as the time from randomization to the first occurrence of disease recurrence or death from any cause. DFS events include: Ipsilateral invasive breast tumor recurrence; Ipsilateral local-regional invasive breast cancer recurrence; Distant recurrence that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer; Contralateral invasive breast cancer; Ipsilateral or contralateral DCIS; Second primary non-breast invasive cancer; Death attributable to any cause. Analysis used Kaplan-Meier estimates where participants with no events at the time of analysis or no post-baseline information were censored.
Time Frame: From randomization up to first disease recurrence or death from any cause (up to 5 years)
Population: ITT population included all randomized participants, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1098 | 1101
months | NA [NA to NA] — Median and 95% CI for DFS were not estimable due to too few events having occurred | NA [NA to NA] — Median and 95% CI for DFS were not estimable due to too few events having occurred

9. Secondary Outcome: Change From Baseline (CFB) in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Patient-reported Function (Role Functioning [Q6, Q7])
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. For the role functioning scale, participant responses to the 2 questions "Q6: Were you limited in doing either your work or daily activities" and "Q7: Were you limited in pursuing your hobbies or other leisure time activities" were scored on a 4-point scale (1=Not at All to 4=Very Much). The scores were linearly transformed on a scale of 0 to 100, with a low score indicating better functioning. Negative change from baseline indicated improvement.
Time Frame: Baseline (Cycle 1 Day 1), Day 1 of Cycles 4, 6, 8, 10, 12, 14 & 16; end of treatment/discontinuation (approximately at Day 351); Follow up: Months 3 to 48 (Total duration is up to 5 years); Cycles 1-5= 28 day cycles; Cycles 6-16: 21 day cycles
Population: Patient-reported outcome (PRO)-evaluable populations included participants in the ITT population with baseline PRO assessment and at least one post-baseline PRO assessment in the EORTC QLQC30. ITT population included all randomized participants, whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1083 | 1088
score on scale
  Baseline | 87.26 (18.92) | 86.43 (19.66)
  CFB: Cycle 4 Day 1: number analyzed (Participants) | 1025 | 1040
  CFB: Cycle 4 Day 1 | -10.88 (25.00) | -10.26 (24.87)
  CFB: Cycle 6 Day 1: number analyzed (Participants) | 938 | 924
  CFB: Cycle 6 Day 1 | -17.31 (29.94) | -16.56 (29.18)
  CFB: Cycle 8 Day 1: number analyzed (Participants) | 902 | 881
  CFB: Cycle 8 Day 1 | -4.58 (23.58) | -4.58 (24.31)
  CFB: Cycle 10 Day 1: number analyzed (Participants) | 898 | 851
  CFB: Cycle 10 Day 1 | -3.77 (23.59) | -3.43 (22.77)
  CFB: Cycle 12 Day 1: number analyzed (Participants) | 869 | 806
  CFB: Cycle 12 Day 1 | -1.53 (22.39) | -1.59 (23.05)
  CFB: Cycle 14 Day 1: number analyzed (Participants) | 830 | 736
  CFB: Cycle 14 Day 1 | -1.02 (21.69) | -0.70 (20.61)
  CFB: Cycle 16 Day 1: number analyzed (Participants) | 628 | 489
  CFB: Cycle 16 Day 1 | -1.09 (23.16) | -0.10 (21.77)
  CFB: Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 896 | 964
  CFB: Study Drug Completion/Early Discontinuation | -2.66 (23.48) | -4.37 (26.12)
  CFB: Follow-up Month 3: number analyzed (Participants) | 845 | 872
  CFB: Follow-up Month 3 | -0.26 (22.62) | -0.40 (23.34)
  CFB: Follow-up Month 6: number analyzed (Participants) | 815 | 818
  CFB: Follow-up Month 6 | 0.20 (24.08) | 0.02 (24.03)
  CFB: Follow-up Month 9: number analyzed (Participants) | 758 | 741
  CFB: Follow-up Month 9 | -0.18 (23.52) | 0.47 (23.35)
  CFB: Follow-up Month 12: number analyzed (Participants) | 677 | 697
  CFB: Follow-up Month 12 | 0.32 (22.42) | 1.22 (21.95)
  CFB: Follow-up Month 18: number analyzed (Participants) | 528 | 548
  CFB: Follow-up Month 18 | -0.47 (24.41) | 1.52 (21.82)
  CFB: Follow-up Month 24: number analyzed (Participants) | 374 | 393
  CFB: Follow-up Month 24 | 0.67 (23.54) | 1.74 (22.28)
  CFB: Follow-up Month 30: number analyzed (Participants) | 223 | 249
  CFB: Follow-up Month 30 | 2.24 (23.36) | 2.01 (24.19)
  CFB: Follow-up Month 36: number analyzed (Participants) | 119 | 130
  CFB: Follow-up Month 36 | 3.08 (23.57) | 4.74 (20.36)
  CFB: Follow-up Month 48: number analyzed (Participants) | 1 | 5
  CFB: Follow-up Month 48 | 0.00 (NA) — The standard deviation was not estimable for one participant. | 13.33 (13.94)

10. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Patient-reported Function (Physical Functioning [Q1-Q5])
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. For the physical functioning scale, participant responses to 5 questions about daily activities (strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves, or using the toilet) were scored on a 4-point scale (1=Not at All to 4=Very Much). The scores were linearly transformed on a scale of 0 to 100, with a high score indicating worst functioning. Negative change from baseline indicated improvement in functioning.
Time Frame: as for outcome 9
Population: PRO-evaluable populations included participants in the ITT population with baseline PRO assessment and at least one post-baseline PRO assessment in the EORTC QLQC30. ITT population included all randomized participants, whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1083 | 1089
score on scale
  Baseline | 89.86 (12.14) | 89.92 (11.57)
  CFB: Cycle 4 Day 1: number analyzed (Participants) | 1025 | 1042
  CFB: Cycle 4 Day 1 | -8.93 (14.97) | -8.69 (14.91)
  CFB: Cycle 6 Day 1: number analyzed (Participants) | 938 | 925
  CFB: Cycle 6 Day 1 | -13.30 (18.63) | -13.55 (18.47)
  CFB: Cycle 8 Day 1: number analyzed (Participants) | 901 | 882
  CFB: Cycle 8 Day 1 | -5.33 (13.79) | -6.42 (14.41)
  CFB: Cycle 10 Day 1: number analyzed (Participants) | 898 | 852
  CFB: Cycle 10 Day 1 | -3.71 (13.28) | -4.42 (13.15)
  CFB: Cycle 12 Day 1: number analyzed (Participants) | 871 | 807
  CFB: Cycle 12 Day 1 | -2.41 (12.87) | -3.42 (12.95)
  CFB: Cycle 14 Day 1: number analyzed (Participants) | 829 | 736
  CFB: Cycle 14 Day 1 | -1.41 (12.87) | -1.92 (12.11)
  CFB: Cycle 16 Day 1: number analyzed (Participants) | 627 | 489
  CFB: Cycle 16 Day 1 | -1.65 (12.78) | -1.82 (12.12)
  CFB:Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 895 | 965
  CFB:Study Drug Completion/Early Discontinuation | -2.56 (13.72) | -4.68 (16.69)
  CFB:Follow-up Month 3: number analyzed (Participants) | 844 | 871
  CFB:Follow-up Month 3 | -1.62 (12.71) | -2.29 (13.47)
  CFB: Follow-up Month 6: number analyzed (Participants) | 815 | 818
  CFB: Follow-up Month 6 | -1.70 (13.46) | -1.96 (13.78)
  CFB: Follow-up Month 9: number analyzed (Participants) | 757 | 741
  CFB: Follow-up Month 9 | -1.55 (13.75) | -1.33 (13.91)
  CFB: Follow-up Month 12: number analyzed (Participants) | 676 | 697
  CFB: Follow-up Month 12 | -1.70 (13.85) | -1.37 (13.39)
  CFB: Follow-up Month 18: number analyzed (Participants) | 527 | 548
  CFB: Follow-up Month 18 | -1.92 (13.60) | -0.91 (13.79)
  CFB: Follow-up Month 24: number analyzed (Participants) | 374 | 392
  CFB: Follow-up Month 24 | -1.37 (13.89) | -0.72 (12.91)
  CFB: Follow-up Month 30: number analyzed (Participants) | 223 | 249
  CFB: Follow-up Month 30 | -1.61 (15.61) | -0.74 (12.72)
  CFB: Follow-up Month 36: number analyzed (Participants) | 119 | 130
  CFB: Follow-up Month 36 | -0.42 (14.40) | 0.82 (13.18)
  CFB: Follow-up Month 48: number analyzed (Participants) | 1 | 5
  CFB: Follow-up Month 48 | -13.33 (NA) — The standard deviation was not estimable for one participant. | -2.67 (3.65)

11. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Global Health Status (GHS) [Q29] and Health-Related Quality of Life (HRQoL) [Q30] Combined Score
Description: The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (Q29:GHS; "How would you rate your overall health during the past week?") and Quality of Life (Q30: QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better outcome. Negative change from Baseline values indicated deterioration in QOL or functioning and positive values indicated improvement.
Time Frame: Baseline (Cycle 1 Day 1), Day 1 of Cycles 4, 6, 8, 10, 12, 14 & 16; end of treatment/discontinuation (approximately 351 days); Follow up: Months 3 to 48 (Total duration is up to 5 years); Cycles 1-5= 28 day cycles; Cycles 6-16: 21 day cycles
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1081 | 1087
score on scale
  Baseline | 76.26 (18.15) | 75.90 (18.52)
  CFB: Cycle 4 Day 1: number analyzed (Participants) | 1022 | 1040
  CFB: Cycle 4 Day 1 | -10.49 (20.25) | -10.02 (19.48)
  CFB: Cycle 6 Day 1: number analyzed (Participants) | 933 | 924
  CFB: Cycle 6 Day 1 | -15.87 (23.83) | -15.68 (22.32)
  CFB: Cycle 8 Day 1: number analyzed (Participants) | 899 | 881
  CFB: Cycle 8 Day 1 | -3.54 (19.72) | -5.09 (18.88)
  CFB: Cycle 10 Day 1: number analyzed (Participants) | 893 | 851
  CFB: Cycle 10 Day 1 | -1.84 (19.57) | -2.82 (18.38)
  CFB: Cycle 12 Day 1: number analyzed (Participants) | 869 | 805
  CFB: Cycle 12 Day 1 | -0.71 (19.41) | -2.31 (18.91)
  CFB: Cycle 14 Day 1: number analyzed (Participants) | 828 | 736
  CFB: Cycle 14 Day 1 | -0.37 (19.04) | -1.25 (18.35)
  CFB: Cycle 16 Day 1: number analyzed (Participants) | 627 | 489
  CFB: Cycle 16 Day 1 | 0.08 (18.56) | -1.30 (18.34)
  CFB:Study Drug Completion/Early Discontinuation: number analyzed (Participants) | 894 | 962
  CFB:Study Drug Completion/Early Discontinuation | -1.56 (20.68) | -4.39 (22.01)
  CFB: Follow-up Month 3: number analyzed (Participants) | 843 | 871
  CFB: Follow-up Month 3 | 1.01 (20.25) | -0.74 (20.50)
  CFB: Follow-up Month 6: number analyzed (Participants) | 813 | 815
  CFB: Follow-up Month 6 | 1.10 (20.23) | -0.90 (20.72)
  CFB: Follow-up Month 9: number analyzed (Participants) | 756 | 740
  CFB: Follow-up Month 9 | 0.62 (20.47) | 0.07 (20.83)
  CFB: Follow-up Month 12: number analyzed (Participants) | 675 | 697
  CFB: Follow-up Month 12 | 1.21 (20.42) | 0.19 (19.84)
  CFB: Follow-up Month 18: number analyzed (Participants) | 526 | 547
  CFB: Follow-up Month 18 | 1.09 (22.18) | 0.47 (20.77)
  CFB: Follow-up Month 24: number analyzed (Participants) | 373 | 390
  CFB: Follow-up Month 24 | 2.32 (22.30) | 0.43 (21.33)
  CFB: Follow-up Month 30: number analyzed (Participants) | 222 | 248
  CFB: Follow-up Month 30 | 1.54 (21.36) | -0.57 (22.43)
  CFB: Follow-up Month 36: number analyzed (Participants) | 117 | 129
  CFB: Follow-up Month 36 | 2.64 (20.95) | 0.58 (23.57)
  CFB: Follow-up Month 48: number analyzed (Participants) | 1 | 4
  CFB: Follow-up Month 48 | 0.00 (NA) — The standard deviation was not estimable for one participant. | 6.25 (31.46)

12. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs are reported based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.
Time Frame: Up to 5 years
Population: Safety Evaluable Population included all participants who received any amount of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1084 | 1093
Participants | 1074 | 1090

13. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Postdose Day 1 of Cycle 1; Predose Day 1 of Cycles 2, 3, and 4; Predose Cycles 6, 10, and 14; Predose Day 2 of Cycle 16; Cycles 1-5= 28-day cycles; Cycles 6-16: 21-day cycles
Population: Pharmacokinetic (PK)-evaluable population included all participants who received any dose of study medication and who have at least one evaluable postbaseline PK sample. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 952
microgram per milliliter (µg/mL)
  Post-dose: Cycle 1 Day 1: number analyzed (Participants) | 853
  Post-dose: Cycle 1 Day 1 | 319 (43.3)
  Pre-dose: Cycle 2 Day 1: number analyzed (Participants) | 854
  Pre-dose: Cycle 2 Day 1 | 153 (85.2)
  Pre-dose: Cycle 3 Day 1: number analyzed (Participants) | 833
  Pre-dose: Cycle 3 Day 1 | 220 (62.0)
  Pre-dose: Cycle 4 Day 1: number analyzed (Participants) | 819
  Pre-dose: Cycle 4 Day 1 | 221 (120.4)
  Pre-dose: Cycle 6: number analyzed (Participants) | 727
  Pre-dose: Cycle 6 | 239 (146.9)
  Pre-dose: Cycle 10: number analyzed (Participants) | 650
  Pre-dose: Cycle 10 | 250 (92.2)
  Pre-dose: Cycle 14: number analyzed (Participants) | 556
  Pre-dose: Cycle 14 | 258 (118.7)
  Pre-dose: Cycle 16 Day 2: number analyzed (Participants) | 2
  Pre-dose: Cycle 16 Day 2 | 355 (29.5)

14. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Baseline evaluable participant= participant with an ADA assay result from a baseline sample(s). Post-baseline evaluable participant= participant with an ADA assay result from at least one postbaseline sample.
Time Frame: Up to 5 years
Population: Safety Evaluable Population included all participants who received any amount of any study drug. Number analyzed at baseline and postbaseline are unique number of participants out of all the assessed participants who may have been ADA positive at that timepoint. Different participants may have contributed data for baseline and postbaseline.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab and Chemotherapy
Number analyzed (Participants) | 1093
percentage of participants
  Baseline: number analyzed (Participants) | 899
  Baseline | 2.1
  Post-baseline: number analyzed (Participants) | 901
  Post-baseline | 11.5

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All-cause Mortality: ITT population population included all randomized participants, whether or not the assigned study treatment was received.; Adverse Events: Safety Evaluable Population included all participants who received any amount of any study drug.
Arm/Group | Chemotherapy | Atezolizumab and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 58/1098 | 72/1101
Serious Adverse Events (participants affected / at risk) | 173/1084 | 280/1093
Other Adverse Events (participants affected / at risk) | 1068/1084 | 1082/1093
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=1084) | Atezolizumab and Chemotherapy (N=1093)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 23 (25) | 29 (35)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (6) | 18 (28)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 3 (4) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 31 (41) | 40 (76)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 6 (6)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 3 (3)
Hypopituitarism (Endocrine disorders) | 0 (0) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 3 (3)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Implant site inflammation (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 4 (4) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (5)
Pyrexia (General disorders) | 10 (10) | 13 (13)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 9 (9)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (3)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 17 (17) | 18 (18)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 6 (7)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 7 (7)
Neutrophil count decreased (Investigations) | 14 (14) | 11 (16)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 6 (6) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 18 (20)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Postoperative care (Surgical and medical procedures) | 0 (0) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=1084) | Atezolizumab and Chemotherapy (N=1093)
Anaemia (Blood and lymphatic system disorders) | 422 (546) | 420 (586)
Leukopenia (Blood and lymphatic system disorders) | 139 (274) | 137 (317)
Neutropenia (Blood and lymphatic system disorders) | 240 (437) | 236 (474)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 62 (65)
Hypothyroidism (Endocrine disorders) | 6 (6) | 161 (173)
Abdominal pain (Gastrointestinal disorders) | 61 (73) | 72 (79)
Abdominal pain upper (Gastrointestinal disorders) | 52 (53) | 79 (92)
Constipation (Gastrointestinal disorders) | 210 (252) | 231 (270)
Diarrhoea (Gastrointestinal disorders) | 188 (260) | 287 (430)
Dyspepsia (Gastrointestinal disorders) | 58 (73) | 65 (71)
Nausea (Gastrointestinal disorders) | 531 (865) | 553 (958)
Stomatitis (Gastrointestinal disorders) | 120 (133) | 143 (166)
Vomiting (Gastrointestinal disorders) | 146 (212) | 177 (242)
Asthenia (General disorders) | 230 (373) | 234 (455)
Fatigue (General disorders) | 268 (348) | 325 (490)
Malaise (General disorders) | 73 (83) | 81 (92)
Oedema peripheral (General disorders) | 76 (84) | 73 (83)
Pyrexia (General disorders) | 105 (126) | 160 (211)
COVID-19 (Infections and infestations) | 34 (34) | 71 (72)
Infusion related reaction (Injury, poisoning and procedural complications) | 70 (95) | 74 (90)
Radiation skin injury (Injury, poisoning and procedural complications) | 13 (13) | 95 (98)
Alanine aminotransferase increased (Investigations) | 240 (319) | 296 (457)
Aspartate aminotransferase increased (Investigations) | 159 (215) | 246 (372)
Blood alkaline phosphatase increased (Investigations) | 38 (43) | 61 (92)
Blood lactate dehydrogenase increased (Investigations) | 57 (106) | 51 (67)
Lymphocyte count decreased (Investigations) | 86 (162) | 113 (214)
Neutrophil count decreased (Investigations) | 254 (473) | 273 (558)
Weight decreased (Investigations) | 27 (30) | 63 (67)
White blood cell count decreased (Investigations) | 196 (392) | 232 (526)
Decreased appetite (Metabolism and nutrition disorders) | 144 (185) | 213 (275)
Hyperglycaemia (Metabolism and nutrition disorders) | 51 (64) | 73 (89)
Arthralgia (Musculoskeletal and connective tissue disorders) | 150 (246) | 218 (333)
Back pain (Musculoskeletal and connective tissue disorders) | 73 (92) | 116 (145)
Bone pain (Musculoskeletal and connective tissue disorders) | 62 (72) | 68 (79)
Myalgia (Musculoskeletal and connective tissue disorders) | 175 (309) | 202 (347)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 50 (58) | 66 (82)
Dizziness (Nervous system disorders) | 58 (68) | 71 (104)
Dysgeusia (Nervous system disorders) | 117 (127) | 116 (129)
Headache (Nervous system disorders) | 135 (178) | 176 (284)
Hypoaesthesia (Nervous system disorders) | 94 (106) | 91 (111)
Neuropathy peripheral (Nervous system disorders) | 151 (179) | 158 (181)
Paraesthesia (Nervous system disorders) | 75 (99) | 72 (117)
Peripheral sensory neuropathy (Nervous system disorders) | 185 (193) | 196 (207)
Insomnia (Psychiatric disorders) | 116 (122) | 140 (158)
Cough (Respiratory, thoracic and mediastinal disorders) | 79 (85) | 132 (158)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 (64) | 84 (105)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 73 (92) | 56 (63)
Alopecia (Skin and subcutaneous tissue disorders) | 715 (733) | 735 (752)
Dry skin (Skin and subcutaneous tissue disorders) | 36 (38) | 55 (57)
Nail discolouration (Skin and subcutaneous tissue disorders) | 99 (108) | 106 (113)
Pruritus (Skin and subcutaneous tissue disorders) | 50 (56) | 127 (160)
Rash (Skin and subcutaneous tissue disorders) | 89 (110) | 167 (200)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 41 (50) | 79 (91)
Hot flush (Vascular disorders) | 50 (52) | 63 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03498716/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03498716/SAP_001.pdf